CLINICAL TRIAL: NCT00187759
Title: A Placebo Controlled, Randomized, and Blinded Study of Antibiotic Treatment of Patients With Uncomplicated Soft Tissue Infection
Brief Title: Placebo Controlled Study of Antibiotic Treatment of Soft Tissue Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS placebo
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Soft Tissue Infections
Keywords: Abscess; Antibitoics; Methicillin-resistant Staphylococcus aureus
MeSH Terms: conditions — Soft Tissue Infections; Abscess | interventions — Cephalexin

INTERVENTIONS:
Drug: cephalexin

SUMMARY:
This study is to determine whether antibiotic therapy is needed for patients with non-life threatening soft tissue infections. Most patients with these soft tissue infections are presently treated with antibiotics. Many of these infections resolve without proper antibiotic treatment. Treatment of patients with antibiotics after surgical drainage of an abscess may not be necessary and indiscriminate use of antibiotics may lead to colonization by drug-resistant organisms. Subsequent infection by drug resistant organisms may limit the choice of antibiotics in more complicated infections. A comparison between antibiotic treatment and no antibiotic treatment in surgically treated, uncomplicated soft tissue infections is needed to address this very important question.

DETAILED DESCRIPTION:
The Integrated Soft Tissue Infection Service (ISIS) Clinic at San Francisco General Hospital treats a large number of patients with soft tissue infections, and our data suggest that antibiotics may be overused for these infections. Most of these infections are treated by surgical drainage of an abscess (77%). When microbiologic cultures were performed, 88% of the abscesses were infected with Staphylococcus aureus (S. aureus), and 55% of the abscesses contained methicillin-resistant Staphylococcus aureus (MRSA). Recently, the high prevalence of MRSA infection has been documented in San Francisco and throughout the country. Presently, most patients are treated with antibiotics after drainage of the abscess. Our retrospective analysis found that 60% of these infections resolved without appropriate antibiotic treatment. These were patients infected with MRSA who were treated with an antibiotic that was not active against that organism. This implies that surgical drainage of these abscesses was probably the important treatment and antibiotic treatment was probably not necessary.

Unnecessary use of antibiotics has adverse consequences. Some patients have allergic reactions to antibiotics. Patients can develop serious gastrointestinal infections from antibiotic use. Antibiotics are costly. But most importantly, overuse of antibiotics may be the significant factor in the spread of antibiotic resistant organisms. The increased prevalence of MRSA has made it extremely difficult to treat patients with appropriate antibiotics in life threatening infections (i.e. bacterial endocarditis, osteomyelitis, and necrotizing soft tissue infections).

The experience in the ISIS Clinic has brought into question our present practice of antibiotic use in patients with surgically managed abscesses. Many surgeons practicing in the ISIS clinic believe that antibiotics have little or no effect on the clinical course of these uncomplicated infections. Elimination of antibiotic use for these uncomplicated infections would certainly simplify care for these patients. It is even possible that decreased antibiotic use may decrease the prevalence of MRSA colonization in this population. However, decreased prevalence of MRSA colonization will not be specifically addressed in this limited study. A randomized, prospective and blinded trial comparing standard antibiotic treatment with no treatment should help determine whether antibiotics are really needed for these infections.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients must have a complicated skin or skin-structure infection that meets disease diagnostic criteria (severity, definition of complicated, and disease).

SEVERITY: Complicated soft tissue infections must be of sufficient severity to anticipate five or more days of antibiotic therapy.

DEFINITION OF COMPLICATED (one or more of the following criteria must be met): Infection requires(ed) significant surgical intervention (such as debridement of devitalized tissue, drainage of abscess, removal of foreign body implicated in infection) at the time of enrollment.

DISEASE: Major Abscess (no open wound). The patient must have all of the following: i) Acute onset within seven days prior to enrollment. ii) Purulent drainage or purulent aspirate. iii) Erythema, induration, or tenderness. iv) Evidence of loculated fluid by physical examination, blind aspiration, or ultrasound that requires intervention (such as aspiration, incision and drainage, excision) at the time of enrollment.

2. A culture must be obtained at the time of enrollment. 3. Patients must be at least 18 years of age. 4. The patient must sign and date a Committee on Human Research-approved informed consent form.

Exclusion Criteria:

1. Any of the following conditions:

   1. Patients unlikely to survive through the treatment period and evaluations.
   2. Conditions such as toxic shock syndrome or toxic-like syndrome (Mandell et al. 2000), shock or hypotension (supine systolic blood pressure <80 mmHg) refractory to fluid or short course pressor challenge (four hours or less) or oliguria (urine output <20 mL/hr) not responsive to fluid challenge.
   3. Incisional wound that extends into visceral compartments.
   4. Suspected or proven contiguous bony or joint involvement.
   5. Malignant otitis externa.
   6. Ischemic ulcers or wounds associated with sever arterial insufficiency or gangrene.
   7. Infection of prosthetic materials or venous catheters that cannot be removed as part of the treatment of the current infection.
   8. Infection of a full-thickness burn wound or burn wound that is >20% total body area.
2. Surgical/nonsurgical debridement of devitalized tissue, removal of prosthetic material, incision and drainage, suture removal, percutaneous aspiration, packing, dressings, or irrigation (including with antibiotics) that cannot be instituted at the time of enrollment.
3. Any known sensitivity to cephalexin.
4. Patients with renal compromise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-11; Study Completion 2005-03

PRIMARY OUTCOMES:
Cure of soft tissue infection.

CONTACTS AND LOCATIONS:
Overall Officials: David M Young, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States